CLINICAL TRIAL: NCT04051190
Title: Effects of Diet-induced Weight Loss Versus Sleeve Gastrectomy and Gastric Bypass on Homeostatic and Hedonic Appetite Markers and Gut Microbiota
Brief Title: Effect of Diet Versus Sleeve Gastrectomy and Gastric Bypass on Appetite
Acronym: DISGAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: St. Olavs Hospital (Other); Namsos Hospital (Other); University of Copenhagen (Other); University of Leeds (Other); Norwegian University of Life Sciences (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019/252
Record Dates: First submitted 2019-08-07; First posted 2019-08-09 (Actual); Last update posted 2023-07-25 (Actual); Status verified 2023-07

CONDITIONS: Obesity
Keywords: diet; bariatric surgery; appetite
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- VLED group (Experimental): Participants will undergo a 10-week VLED.
  Interventions: Dietary Supplement: VLED group
- Sleeve Gastrectomy group (Experimental): Participants will undergo standard clinical practice prior to surgery.
  Interventions: Dietary Supplement: VLED group; Procedure: Sleeve Gastrectomy group
- Gatric Bypass group (Experimental): Participants will undergo standard clinical practice prior to surgery.
  Interventions: Dietary Supplement: VLED group; Procedure: Gastric Bypass group

INTERVENTIONS:
Dietary Supplement: VLED group — 10-week weight loss period with total meal replacement, consisting of 750 kcal/day. Measurements will be taken at baseline (before diet start), 10 weeks after intervention start (Wk11), and at 1 year.
  Other Names: very-low-energy-diet
Procedure: Sleeve Gastrectomy group — Standard clinical practice with 2-week diet consisting of 750 kcal/day prior to surgery. The pre- and post-surgical diet of this group will be matched with the VLED group in macro- and micronutrient composition. Measurements will be taken at baseline (before diet start), 10 weeks after intervention start (Wk11), and 1 year after surgery (sleeve gastrectomy)
  Arms: Sleeve Gastrectomy group
Procedure: Gastric Bypass group — Standard clinical practice with 2-week diet consisting of 750 kcal/day prior to surgery. The pre- and post-surgical diet of this group will be matched with the VLED group in macro- and micronutrient composition. Measurements will be taken at baseline (before diet start), 10 weeks after intervention start (Wk11), and 1 year after surgery (gastric bypass)
  Arms: Gatric Bypass group

SUMMARY:
The biggest challenge in obesity management is maintaining weight loss in the long-term. Currently, bariatric surgery is the most effective treatment, leading to sustained weight loss that is not yet achievable with lifestyle intervention (e.g. diet). The reasons behind its success is still not clearly understood, but beneficial changes in the homeostatic and hedonic appetite systems (the two major physiological regulators of appetite), along with the microbiome (known to have a mediatory effect on appetite) have been shown to occur after bariatric surgery. These alterations are in opposition to what is seen after diet-induced weight loss. Today, the component of appetite regulation that drives bariatric surgeys' long-term success is still unknown. By comparing a lifestyle and surgical intervention in parallel, the investigators can observe the impact of a similar magnitude of weight loss on these three domains of appetite regulation simultaneously, thereby illuminating the mechanisms behind bariatric surgerys' success.

ELIGIBILITY:
Inclusion Criteria:

* scheduled for bariatric surgery
* patient in obesity clinic
* Body mass index (BMI) 35-55

Exclusion Criteria:

* Currently taking medication known to affect energy metabolism or appetite
* Current cancer diagnosis
* Substance abuse
* Enrolled in another obesity treatment
* Eating disorders
* pre-existing endocrine disorders (e.g. diabetes) will not be excluded, but final analysis will controlled for these conditions

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2019-09-02 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Postprandial blood plasma concentration of Glucagon-like peptide-1 (GLP-1, satiety hormone) | Week 11
  Blood samples will be collected at fasting, and then every 30 minutes after a standardized test meal up to 150 minutes. A radioimmunoassay method will be used to measure the concentration of total GLP-1. This method measures antigen concentrations by the use of antibodies.

CONTACTS AND LOCATIONS:
Overall Officials: Catia Martins, PhD, Principal Investigator — Norwegian University of Science and Technology
Locations (2):
- Norway (2):
  - Namsos Hospital, Namsos
  - St. Olavs Hospital, Trondheim

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Finn A, Cedillo Y, Aukan M, Gower B, Martins C. Glucose-Dependent Insulinotropic Polypeptide and Glucagon After Weight Loss Induced by Diet or Bariatric Surgery. Obesity (Silver Spring). 2025 Dec;33(12):2277-2288. doi: 10.1002/oby.70049. Epub 2025 Sep 29. PMID 41024443
- [Derived] Aukan MI, Rehfeld JF, Holst JJ, Martins C. Plasma concentration of gastrointestinal hormones and subjective appetite ratings after diet or bariatric surgery: 1-year results from the DISGAP study. Int J Obes (Lond). 2025 Feb;49(2):306-314. doi: 10.1038/s41366-024-01658-5. Epub 2024 Nov 21. PMID 39572763
- [Derived] Martins C, Aukan MI, De Luca M. Lower levels of plasma syndecan-4 are associated with loss of body weight and fat-free mass after bariatric surgery. BMC Res Notes. 2024 Jun 15;17(1):164. doi: 10.1186/s13104-024-06822-8. PMID 38879520
- [Derived] Martins C, Nymo S, Aukan MI, Roekenes JA, Coutinho SR, Hunter GR, Gower BA. Association between ss-Hydroxybutyrate Plasma Concentrations after Hypocaloric Ketogenic Diets and Changes in Body Composition. J Nutr. 2023 Jul;153(7):1944-1949. doi: 10.1016/j.tjnut.2023.05.010. Epub 2023 May 12. PMID 37182692
- [Derived] Aukan MI, Brandsaeter IO, Skarvold S, Finlayson G, Nymo S, Coutinho S, Martins C. Changes in hedonic hunger and food reward after a similar weight loss induced by a very low-energy diet or bariatric surgery. Obesity (Silver Spring). 2022 Oct;30(10):1963-1972. doi: 10.1002/oby.23535. Epub 2022 Aug 31. PMID 36046953
- [Derived] Nymo S, Lundanes J, Aukan M, Sandvik J, Johnsen G, Graeslie H, Larsson I, Martins C. Diet and physical activity are associated with suboptimal weight loss and weight regain 10-15 years after Roux-en-Y gastric bypass: A cross-sectional study. Obes Res Clin Pract. 2022 Mar-Apr;16(2):163-169. doi: 10.1016/j.orcp.2022.03.006. Epub 2022 Apr 4. PMID 35393266